CLINICAL TRIAL: NCT02942485
Title: Treatment of Giardia Lamblia Infections in Children: Randomized Open-labeled Trial Comparing Rectal Metronidazole With Oral Tinidazole
Brief Title: Treatment of Giardia Lamblia Infections in Children
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Extremely slow enrollment
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Svetlana Kostjukovits, MD, Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PGLIT2016
Record Dates: First submitted 2016-10-19; First posted 2016-10-24 (Estimated); Results first posted 2020-11-18 (Actual); Last update posted 2020-11-18 (Actual); Status verified 2020-11

CONDITIONS: GIARDIASIS
MeSH Terms: conditions — Giardiasis | interventions — Metronidazole; Tinidazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Metronidazole (Experimental): Patients will be given rectal metronidazole (Flagyl) 500 mg/dose for children weighing 10-14,9 kg, 1000 mg/dose for those weighing 15-29,9 kg and 1500 mg/dose for those weighing 30-44,9 kg. Suppositories will not be halved. Patients will be given 1 dose/day for 3 days.
  Interventions: Drug: Metronidazole
- Tinidazole (Active Comparator): Patients will be treated with a standard regimen of oral tinidazole (Fasigyn) at a single dose of 50 mg/kg, maximum 2 g/dose
  Interventions: Drug: Tinidazole

INTERVENTIONS:
Drug: Metronidazole — P/r suppositories
  Other Names: Flagyl
  Arms: Metronidazole
Drug: Tinidazole — P/o tablets
  Other Names: Fasigyn
  Arms: Tinidazole

SUMMARY:
This study investigates the efficacy and safety of rectally administered metronidazole for pediatric Giardia lamblia infection, as well as the acceptance of this treatment regimen by patients/caregivers. The investigators hypothesize that rectal metronidazole is non-inferior to single-dose of oral tinidazole and will cure at least 72% of patients, a well as will be tolerated as good as tinidazole.

DETAILED DESCRIPTION:
Approximately 180 children (age 6 months to 10 years) whose clinical symptoms could be explained by giardiasis and whose fecal samples will test positive for the presence of G.lamblia in Uusimaa laboratory (HUSLAB) will be recruited.

The study will be performed as an open-label trial. Patients will be randomized during primary visits alternately into two groups by random allocation to receive either of the two study drugs.

Patients from group 1 will be treated with a standard regimen of oral tinidazole (Fasigyn) at a single dose of 50 mg/kg, maximum 2 g/dose. Patients from group 2 will be given rectal metronidazole (Flagyl) 500 mg/dose for children weighing 10-14,9 kg, 1000 mg/dose for those weighing 15-29,9 kg and 1500 mg/dose for those weighing 30-44,9 kg. Suppositories will not be halved. Patients will be given 1 dose/day for 3 days. The first dose of metronidazole will be administered during the primary clinical visit and 2 additional doses will be provided to the parents for home administration.

Fecal samples will be collected from the study patients on day 7-10 post-treatment and will be analyzed in HUSLAB for the presence of G.lamblia antigen by enzyme immunoassay (EIA). Early collection of samples on day 7-10 will help to avoid the risk of tests being positive due to reinfection.

If any of the patients will not clear the infection by day 10, he/she will be invited to a second visit and re-treated. Patients from group 1 will be re-treated by rectal metronidazole and patients from group 2 by oral tinidazole, thus performing a cross-over. Follow-up stool samples will be collected.

Criteria for clinical cure will be resolution of symptoms by day 10 and microbiological cure will be defined as negative G.lamblia antigen test from fecal samples collected on day 7-10 post-treatment.

ELIGIBILITY:
Inclusion Criteria:

* clinical symptoms could be explained by giardiasis AND
* fecal samples will test positive for the presence of G.lamblia in Uusimaa laboratory (HUSLAB)

Exclusion Criteria:

* age <6 mo or >10 years
* weight <9.5 kg
* the absence of symptoms
* co-infection with another pathogen, which may cause giardiasis-like symptoms

Ages: 6 Months to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 8 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital, HYKS, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: Yes

RESULTS

PARTICIPANT FLOW:
Recruitment Details: There were no cross-over patients.
Period: Overall Study
Arm/Group | Metronidazole | Tinidazole
Started | 7 | 1
Completed | 6 | 1
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Metronidazole | Tinidazole | Total
Number analyzed (Participants) | 7 | 1 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 7 | 1 | 8
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 6 | 1 | 7
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Clinical Recovery
Description: Clinical recovery was defined as the resolution of symptoms by day 10 post-treatment, assessed using a structured questionnaire by interviewing the parents/caregivers.
Time Frame: 10 days
Population: 3 participants in the "Metronidazole" and 1 participant "Tinidazole" Arm/Group were asymptomatic and the main primary outcome (clinical cure) could not be assessed
Measure: Count of Participants; unit: Participants
Arm/Group | Metronidazole | Tinidazole
Number analyzed (Participants) | 4 | 0
Participants | 4 | 0

2. Secondary Outcome: Number of Participants With Side-effects
Description: Will be assessed using structured questionnaire by interviewing parents/caregivers.
Time Frame: 10 days
Measure: Count of Participants; unit: Participants
Arm/Group | Metronidazole | Tinidazole
Number analyzed (Participants) | 7 | 1
Participants | 1 | 0

3. Secondary Outcome: Number of Participants With Negative G.Lamblia Antigen Test
Description: Microbiological recovery was defined as negative G.lamblia antigen test from fecal samples collected on day 10 post-treatment.
Time Frame: 10 days
Measure: Count of Participants; unit: Participants
Arm/Group | Metronidazole | Tinidazole
Number analyzed (Participants) | 5 | 1
Participants | 5 | 1

ADVERSE EVENTS:
Time Frame: 1 month
Description: All healthy children
Arm/Group | Metronidazole | Tinidazole
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/1
Other Adverse Events (participants affected / at risk) | 1/7 | 0/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metronidazole (N=7) | Tinidazole (N=1)
diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) — Single episode of loose stools after the third dose of rectal metronidazole

LIMITATIONS AND CAVEATS:
The study was terminated due to the extremely slow patient enrollment: eight patients only have been referred and recruited during the two-year period. 6/8 patients fulﬁlled one or more of the exclusion criteria.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2016-09-01): https://cdn.clinicaltrials.gov/large-docs/85/NCT02942485/Prot_000.pdf